CLINICAL TRIAL: NCT00394238
Title: Non Alcoholic Fatty Liver Disease in Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Other Study IDs: 20174CTIL
Record Dates: First submitted 2006-10-29; First posted 2006-10-31 (Estimated); Last update posted 2006-10-31 (Estimated); Status verified 2006-07

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Procedure: Ultrasonographic imaging

SUMMARY:
Rheumatoid arthritis is a chronic inflammatory systemic disease. It has a worldwide distribution and can affect all age group. The peak incidence is between fourth and sixth decade. It is more prevalent in women, and it's prevalence in the general population in North America is between 0.2-1.5%. The etiology of RA is unknown, although clusters of the disease in families and high concordance in mono-zydotic twins support genetic predisposition. The prevalence of fatty liver disease in patients with rheumatoid arthritis is currently unknown. We wish to study the link between the two conditions by performing a son graphic imaging of the liver in a cohort of RA patients. If indeed a high prevalence of NAFLD will be found in the RA patients, further support will be landed for the link between inflammation and fatty liver disease. These findings may also have implications regarding the management and follow up of RA patients.

The validity of sonographic imaging for detection of fatty liver diseases is currently accepted: On ultrasonographic, fatty infiltration of the liver produces a diffuse increase in echogenicity as compared with that of the kidneys. Ultrasonography has a sensitivity of 89% and a specificity of 93% in detecting steatosis and sensitivity and specificity of 77% and 89% respectively in detecting increase fibrosis.

In view of all the above data, we expected to find higher prevalence of fatty liver in the patients with higher inflammation markers compare with patients with lower markers.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis

Exclusion Criteria:

* Age below 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2006-11; Study Completion 2008-10

CONTACTS AND LOCATIONS:
Overall Officials: Michal Mates, MD, Principal Investigator — Shaare Zedek Medical Center Jerusalem
Locations (1):
- Rheumatoid Clinic, Jerusalem, Israel